CLINICAL TRIAL: NCT05861167
Title: Efficacy and Safety of Selective Intensive Induction Therapy Based on Ustekinumab Clinical Decision-making Tools in Patients With Crohn's Disease: A Multicenter, Prospective, Randomized, Controlled Study（SIIT-CD Study）
Brief Title: SIIT Based on UST CDST in Patients With CD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Gao, Sixth Affiliated Hospital, Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZSLYEC-353
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIIT group (Experimental)
  Interventions: Biological: selective intensive induction therapy based on ustekinumab clinical decision-making tools
- Non-intensive induction therapy group (No Intervention)

INTERVENTIONS:
Biological: selective intensive induction therapy based on ustekinumab clinical decision-making tools — At week 0 and week 8, UST was induced intravenously twice (stratified according to body weight, see instructions for dosage), and at the third time, intravenous or standard subcutaneous injection regimen was used according to CRP standard
  Arms: SIIT group

SUMMARY:
ustekinumab (UST) can effectively induce and maintain clinical remission and mucosal healing of Crohn's disease (CD), but some patients still have poor response. Dose optimization is an effective way to improve the response rate of UST, and re-intravenous induction is a common way of optimization. For patients with secondary loss of response, about half of the patients can re-respond after dose optimization. We plan to use CDST-UST to stratify the response level of patients before treatment, select patients with poor response, and initially give multiple intravenous therapy as an intensive induction therapy strategy, so as to improve the response rate of these patients and achieve individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CD;
* Active period; Age 18-75 years old;
* UST-CDST scores were used to treat patients with moderate and low responsive activity

Exclusion Criteria:

* Subjects had undergone extensive colectomy, subtotal colectomy, or total colectomy; The subject currently has ileostomy and colostomy; Patients with significant liver, kidney, endocrine, respiratory, neurological or cardiovascular diseases; Patients with fibrous stenosis and prestenosis dilatation; Contraindications of UST as documented in other specifications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in clinical response rate at week 24 between intensive induction regimen and standard induction regimen | week 24
  Difference in clinical response rate at week 24 between intensive induction regimen and standard induction regimen

CONTACTS AND LOCATIONS:
Locations (1):
- SixthSunYetSen, Guangzhou, 省/直辖市, China

IPD SHARING:
Plan to Share IPD: Undecided